CLINICAL TRIAL: NCT04614519
Title: Appendectomy by Low Impact Laparoscopy vs Routine Laparoscopy : a Randomized Prospective Monocentric Trial
Acronym: LIL-APP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-AOI-02
Record Dates: First submitted 2020-10-29; First posted 2020-11-04 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Appendicitis; Appendectomy
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional group (Active Comparator): Insufflation pressure at 12mmHg and conventional instrumentation
  Interventions: Procedure: Conventional group
- Low impact laparoscopy group (Experimental): Insufflation pressure at 7mmHg and micro-laparoscopy instrumentation
  Interventions: Procedure: Low impact laparoscopy group

INTERVENTIONS:
Procedure: Conventional group — Insufflation pressure at 12mmHg and conventional instrumentation
  Arms: Conventional group
Procedure: Low impact laparoscopy group — Insufflation pressure at 7mmHg and micro-laparoscopy instrumentation
  Arms: Low impact laparoscopy group

SUMMARY:
Introduction: Surgery performed under low insufflation pressure combined with micro-laparoscopy (incisions 4X smaller than incisions in conventional laparoscopy) is called "low impact laparoscopy" or LIL. It significantly reduces postoperative pain and reduces the average length of stay.

This technique, currently underdeveloped has never been evaluated in the literature for appendectomy.

Main objective of the study: to obtain a reduction in postoperative pain when using the low-impact laparoscopy technique for appendectomies.

Secondary objectives: to study the feasibility of LIL in appendectomies, to obtain a reduction in the average length of stay, a reduction in the consumption of analgesics, a reduction in costs, and a more rapid resumption of activities.

Material and methods :

This is a prospective, single-center, double-blind study. The inclusion criterion is the presence of acute uncomplicated appendicitis. The number of subjects to be included in each group is evaluated at 25. The subjects are divided into two groups preoperatively:

* Conventional group: insufflation pressure at 12mmHg and conventional instrumentation
* LIL group: insufflation pressure at 7mmHg and micro-laparoscopy instrumentation.

Identical dressings are put in place at the end of the procedure in order to hide from the patient the protocol in which he was included.

Pain assessment is recorded daily during the first postoperative week. The consumption of analgesics is also recorded. Then on the 7th day, 15th day and 30th postoperative day. During hospitalization, readings are taken by the nurse. At home, the data is entered by the patient via the Link4Life smartphone application.

Conclusion: LIL applied to appendectomy has never been evaluated in the literature. It would allow a reduction in postoperative pain, the average length of stay for patients as well as improved rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

- Patients with acute appendicitis uncomplicated by computed tomography with injection of contrast product

Exclusion Criteria:

* coagulopathy or thrombopathy
* arguments for a complicated appendicitis: fever> 38.5 ° C, hyperleucytosis> 15,000, CRP> 100, presence of an intraperitoneal abscess, a plastron, a fluid effusion of medium or great abundance or '' a pneumoperitoneum on the CT scan
* History of abdominal surgery by laparotomy
* Obese patients (BMI> 30kg / m2)
* minor patients
* patients without health insurance
* pregnant patient
* patient incarcerated or in detention
* patient under guardianship or curatorship
* rapid sequence induction with the use of ketamine

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-01-12 (Actual); Primary Completion 2022-07-22 (Actual); Study Completion 2022-07-22 (Actual)

PRIMARY OUTCOMES:
Post-operative pain decrease with low-impact laparoscopy | 30 days
  Decrease of 2 points on a numerical pain scale of 0 to 10 in the LIL group compared to the conventional group.

SECONDARY OUTCOMES:
Feasibility of Low Impact Laparoscopy in appendectomies | 30 days
  Possibility of performing at least 80% of LIL procedures without conversion to conventional laparoscopy
Reduction in the average length of stay | 30 days
  Obtain a 10% reduction in the average length of stay between the 2 groups
Decrease of opioids consumption | 30 days
  Obtain a 10% reduction in the consumption of level 2 and 3 perioperative analgesics
Cost reduction in the LIL group | 30 days
  Equivalent operating time in the 2 groups
Faster resumption of activities | 30 days
  Lower costs in the LIL group compared to the conventional group

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nice, Nice, France

REFERENCES:
- [Derived] Etienne JH, Salucki B, Gridel V, Orban JC, Baque P, Massalou D. Low-Impact Laparoscopy vs Conventional Laparoscopy for Appendectomy: A Prospective Randomized Trial. J Am Coll Surg. 2023 Oct 1;237(4):622-631. doi: 10.1097/XCS.0000000000000795. Epub 2023 Jun 29. PMID 37382370